CLINICAL TRIAL: NCT02546401
Title: Comparison of Injection of an Analogue Bolus of Insulin Before or After the Meal in Type 1 Diabetic Patients Treated With Insulin Pump.
Brief Title: Comparison of Insulin's Injection Before or After the Meal in Type 1 Diabetic Patients Treated With Insulin Pump
Acronym: BOLUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RB 15-027; 2015-000915-42 (EudraCT Number)
Record Dates: First submitted 2015-09-09; First posted 2015-09-10 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2016-04

CONDITIONS: Diabetes Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; NOP-bolus regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Patients will perform their bolus for 2 weeks before meals (BE) and for 2 weeks after meals (AF).
  Intervention: drug (insulin Aspart)
  Interventions: Drug: Insulin Aspart
- Group 2 (Experimental): Patients will perform their bolus for 2 weeks after meals (AF) and for 2 weeks before meals (BE).
  Intervention: drug (insulin Aspart)
  Interventions: Drug: Insulin Aspart

INTERVENTIONS:
Drug: Insulin Aspart — Injection of Insulin Aspart before or after meals
  Other Names: Bolus

SUMMARY:
The current study focuses on terms of use of Insulin Aspart, fast analogue of human insulin and commonly used in the treatment of type 1 diabetes, where it obtained the marketing authorization for this indication. In the patient who have an insulin pump, insulin Aspart is given daily like a pre-prandial bolus (just before the meal). However, many patients perform their bolus after the meal. However this insulin administration modality is not clearly studied in the literature.

DETAILED DESCRIPTION:
The functional insulin therapy is a method for adjusting insulin doses which tends to mimic the physiology, especially when food intake with proportional dose calculation to the amount of carbohydrates ingested by the use of ratios. This method of adaptation, increasingly used in France, is an extension in the use of subcutaneous insulin pump with a more precise determination of bolus doses with meals, and use of aids dose calculations (assistant wizard for instance). In practice every day, some patients perform their bolus immediately after eating, not just before, allowing them to know exactly the amount of ingested carbohydrates and not the one provided in advance.

This study is very interesting because it allows to compare the injection of an analogous bolus of fast insulin before and after the meal.

ELIGIBILITY:
Inclusion Criteria:

* Major patients with type 1 diabetes treated with insulin pump.

Exclusion Criteria:

* Unbalanced diabetes,
* Ongoing pregnancy known,
* Gastrointestinal neuropathy known,
* Chronic medical illness and psychiatric

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) of glycemia | During 14 days
  Area Under Curve (AUC) recording blood glucose performed continuously over 14 days, with baseline to 1,40g/L (in order not to consider hypoglycemia)

SECONDARY OUTCOMES:
Mean Amplitude of Glycemic excursions (MAGE) = measure of glycemia instability | During 14 days
Area Under Curve (AUC) during 4H after a high-fat meal | 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thuillier P, Sonnet E, Alavi Z, Roudaut N, Nowak E, Dion A, Kerlan V. Comparison between preprandial vs. postprandial insulin aspart in patients with type 1 diabetes on insulin pump and real-time continuous glucose monitoring. Diabetes Metab Res Rev. 2018 Sep;34(6):e3019. doi: 10.1002/dmrr.3019. Epub 2018 Jun 1. PMID 29749032